CLINICAL TRIAL: NCT04317313
Title: Synergistic Effect of 18F-FDG PET Radiomics and International Prognostic Index on Outcome Prediction in Diffuse Large B-cell Lymphoma
Brief Title: 18F-FDG PET Radiomics of Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-350
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: PET; Diffuse large B-cell lymphoma; Prognosis; Radiomics;
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FDG PET radiomic feature evaluation — A total of 1245 radiomic features will be calculated and extracted from baseline FDG PET scans. These features include shape features, first order features, textural features and wavelet features.
  In the second part, based on the results of least absolute shrinkage and selection operator Cox regression algorithm, the most significant radiomic features will be selected to construct the radiomic signature.

SUMMARY:
This study aims to investigate the prognostic value of 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) radiomics in diffuse large B-cell lymphoma (DLBCL) and its additional value to the International Prognostic Index (IPI).

DETAILED DESCRIPTION:
Several studies have shown that 18F-FDG PET radiomics is predictive of survival in DLBCL. However, to the best of the investigator's knowledge, a multi-feature radiomic signature for prognosis assessment of DLBCL has not yet been described. Furthermore, it remains unclear whether PET-based radiomics could add more prognostic values to the IPI in DLBCL.

This study aims to develop 18F-FDG PET radiomic signature, and investigate whether the radiomic signature could improve the prognostic value of the IPI score in predicting progression-free survival (PFS) and overall survival (OS) in DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically confirmed diffuse large B-cell lymphoma (DLBCL);
2. Over 18 years old when diagnosed;
3. Have undergone pre-treatment 18F-FDG PET/CT;
4. Have been initially treated with the combination of rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone (R-CHOP) or R-EPOCH (etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin).

Exclusion Criteria:

1. Have primary central nervous system (CNS) lymphoma or second primary cancer;
2. Have undergone surgical resection;
3. With an incomplete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population of this retrospective study is patients with DLBCL who have undergone pre-treatment 18F-FDG PET/CT prior to the R-CHOP or R-EPOCH chemotherapy. The study will assess the relationships between PET-derived radiomic features with the patient outcome data.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Tian, M.D., Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Chen L, Jiang H, He X, Feng L, Ni M, Ma M, Wang J, Zhang T, Wu S, Zhou R, Jin C, Zhang K, Qian W, Chen Z, Zhuo C, Zhang H, Tian M. A novel analytic approach for outcome prediction in diffuse large B-cell lymphoma by [18F]FDG PET/CT. Eur J Nucl Med Mol Imaging. 2022 Mar;49(4):1298-1310. doi: 10.1007/s00259-021-05572-0. Epub 2021 Oct 15. PMID 34651227

RESULTS

PARTICIPANT FLOW:
Groups:
- Training Cohort: Patients diagnosed between July 2013 and March 2017. All patients underwent pre-treatment 18F-FDG PET/CT. PET/CT images were acquired on a Biograph mCT scanner (Siemens Healthcare, Germany) 60-70 min after intravenous injection of 18F-FDG (3.7 MBq/kg).
- Validation Cohort: Patients diagnosed between April 2017 and July 2019. All patients underwent pre-treatment 18F-FDG PET/CT. PET/CT images were acquired on a Biograph mCT scanner (Siemens Healthcare, Germany) 60-70 min after intravenous injection of 18F-FDG (3.7 MBq/kg).
Period: Overall Study
Arm/Group | Training Cohort | Validation Cohort
Started | 100 | 52
Completed | 100 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Training Cohort: Patients diagnosed between July 2013 and March 2017
- Validation Cohort: Patients diagnosed between April 2017 and July 2019
- Total: Total of all reporting groups
Arm/Group | Training Cohort | Validation Cohort | Total
Number analyzed (Participants) | 100 | 52 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (14.6) | 59.4 (15.7) | 58.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 24 | 76
  Male | 48 | 28 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 100 | 52 | 152
lactate dehydrogenase [Count of Participants; unit: Participants] — Normal: 190-245 U/L; Elevated: > 245 U/L
  Participants
    Normal | 45 | 21 | 66
    Elevated | 55 | 31 | 86
β2-microglobulin [Count of Participants; unit: Participants] — Normal: 1.0 - 3.0 μg/L; Elevated: > 3.0 μg/L
  Participants
    Normal | 67 | 31 | 98
    Elevated | 33 | 21 | 54
Ann Arbor stage [Count of Participants; unit: Participants] — Ann Arbor stage was evaluated based on the Lugano classification. Stage I: only one node or a group of adjacent nodes involved. Stage II: two or more nodal groups on the same side of the diaphragm. Stage III: nodes on both sides of the diaphragm, or nodes above the diaphragm with spleen involvement. Stage IV: additional noncontiguous extralymphatic involvement. Stage I/II were classified as limited stage (with better prognosis), while stage III/IV were defined as advanced stage (with worse prognosis).
  Participants
    Ⅰ-Ⅱ | 38 | 15 | 53
    Ⅲ-Ⅳ | 62 | 37 | 99
Performance status [Count of Participants; unit: Participants] — Performance status was evaluated according to the Eastern Cooperative Oncology Group (ECOG) criteria.
  Score 0: Fully active, able to carry on all pre-disease performance without restriction; Score 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Score 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; Score 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; Score 4: Completely disabled.
  Participants
    < 2 | 76 | 32 | 108
    ≥ 2 | 24 | 20 | 44
B symptoms [Count of Participants; unit: Participants] — The B symptoms were defined as the occurrence of one or more of three symptoms: weight loss (>10% over 6 months), heavy night sweats and fever (>38°C).
  Participants
    Yes | 28 | 20 | 48
    No | 72 | 32 | 104
Extranodal sites [Count of Participants; unit: Participants] — Extranodal sites included the bone marrow, gastrointestinal tract, liver, lung, central nervous system, and other sites. The numbers of extranodal disease sites were recorded as 0, 1, or more than 1.
  Participants
    < 2 | 71 | 30 | 101
    ≥ 2 | 29 | 22 | 51
International Prognostic Index [Count of Participants; unit: Participants] — The International Prognostic Index was defined according to the number of the following risk factors: elevated LDH, age >60 years, ECOG performance score ≥2, involvement of more than one extranodal site, and Ann Arbor stage III/IV.
  Score 0/1: Low risk; Score 2: Low-intermediate risk; Score 3: High-intermediate risk; Score 4: High risk
  Participants
    ≤ 2 | 54 | 30 | 84
    > 2 | 46 | 22 | 68
Cell of origin [Count of Participants; unit: Participants]
  germinal center B-cell like | 28 | 14 | 42
  non-germinal center B-cell like | 72 | 38 | 110
Treatment [Count of Participants; unit: Participants]
  Chemotherapy alone | 72 | 41 | 113
  Chemotherapy + radiotherapy | 25 | 10 | 35
  Chemotherapy + autologous stem cell transplantation | 3 | 1 | 4
Chemotherapy regimens [Count of Participants; unit: Participants] — 1. R-CHOP: rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone;
  2. R-EPOCH: rituximab, etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin
  Participants
    R-CHOP | 95 | 48 | 143
    R-EPOCH | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: the period from the initial diagnosis to the death from any cause
Time Frame: From date of the initial diagnosis until the date of death from any cause, whichever came first, up to 8 years
Measure: Median (Full Range); unit: months
Arm/Group | Training Cohort | Validation Cohort
Number analyzed (Participants) | 100 | 52
months | 56 [4 to 96] | 29 [4.5 to 50]

2. Primary Outcome: Progression-free Survival
Description: the period from the initial diagnosis to the progression, relapse or death from any cause
Time Frame: From date of the initial diagnosis until the date of first documented progression, relapse or death from any cause, whichever came first, up to 8 years
Measure: Median (Full Range); unit: months
Arm/Group | Training Cohort | Validation Cohort
Number analyzed (Participants) | 100 | 52
months | 52.5 [4 to 96] | 28 [4 to 50]

ADVERSE EVENTS:
Time Frame: From patient diagnosis to the end of the study, up to 1 year
Arm/Group | Training Cohort | Validation Cohort
All-Cause Mortality (participants affected / at risk) | 27/100 | 14/52
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/52
Other Adverse Events (participants affected / at risk) | 0/100 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT04317313/Prot_SAP_001.pdf